CLINICAL TRIAL: NCT04662892
Title: A Prospective Observational Registry Study for Real-World Outcome Analysis to Estimate the Incidence of FN Among Subjects Who Are at High Risk for FN, Have Non-myeloid Malignancies, and Are Receiving Udenyca for Prophylaxis of FN
Brief Title: An Analysis to Estimate Febrile Neutropenia (FN) in Patients Receiving Udenyca
Acronym: POEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Community Clinical Oncology Research Network, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: POEM v1.0
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Febrile Neutropenia; Non-myeloid Malignancy
MeSH Terms: conditions — Febrile Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Pegfilgrastim-Cbqv — Date, Dose, and cycle for subjects who received Udenyca will be recorded. Other FN prophylaxis such as Neulasta, or other pegfilgrastim biosimilars will be collected.
  Other Names: Neulasta; pegfilgrastim biosimilar

SUMMARY:
This is a multicenter, prospective, observational cohort registry in subjects receiving myelosuppressive chemotherapy for a non-myeloid malignancy who are considered to be at high risk for developing febrile neutropenia (FN).

DETAILED DESCRIPTION:
Little is known about the real-world risk of febrile neutropenia (FN) among subjects receiving Udenyca. Udenyca was approved due to the totality of evidence under the new Food and Drug Administration (FDA) pathway 351 (k), which met all the endpoints of pharmacokinetic (PK), pharmacodynamic (PD) and immunogenicity in healthy volunteers. Udenyca is the only pegfilgrastim that has not been studied in actual patient cohorts; it has only been studied in healthy volunteers. This prospective observational cohort study is designed to estimate the risk of FN among subjects who 1) are at high risk for FN while receiving myelosuppressive chemotherapy in a real-world outcomes setting and 2) receive Udenyca for FN prophylaxis with each cycle of highly myelotoxic chemotherapy.

Study Plans: After signing the informed consent form, data collection will start at visit 1/cycle 1 (screening/enrollment [day 1]); subjects who received chemotherapy up to 1 week prior to enrollment are eligible to participate in the study.

Visit 1/cycle 1 is to coincide with day 1 (± 7 days) of the subjects' chemotherapy treatment; data collection should start at day 1/visit 1/cycle 1 of chemotherapy. Entries will be recorded during a subject's medical chart review to obtain information on demographic factors, malignancy characteristics (e.g., malignancy histology, date of initial malignancy diagnosis, stage at diagnosis, current malignancy stage, any previous cancer therapy [radiation, surgery, or chemotherapy]), relevant comorbidities, laboratory data, and relevant concomitant therapies.

Subjects' socio-demographic and clinical characteristics will be collected on the date of enrollment and include age, sex, geographic region, health plan information, socioeconomic status (employment status), body surface area, and tobacco use.

Detailed clinical information and laboratory information will be collected, including subjects' medical and treatment history, comorbid conditions, and history of any other malignancies (as well as any treatment received for these other malignancies). Additionally, subject Eastern Cooperative Oncology Group (ECOG) Performance Status, relevant concomitant medications, and any adverse events that occur throughout the study will be recorded.

Subjects will be followed from study enrollment (Cycle 1, Visit 1) throughout the end of their treatment cycle or until the earliest of loss to follow-up, withdrawal of consent, death, end of study (EOS), discontinuation of chemotherapy regimen prior to 4 cycles, or termination of study by the sponsor.

The study data will be captured using the electronic case report form (eCRF), which will contain information collected directly about the subjects and their treatment/outcomes from the healthcare study research personnel. Data will be entered into the eCRF by research coordinators at the individual sites. The data to be entered into the eCRF will be obtained from paper or electronic medical records depending on the technology used by individual sites. The short form health survey SF-12 Health-related Quality of Life (HRQoL) instrument will be used for HRQoL outcomes.

A data management plan will be created and will describe all functions, processes, and specifications for data collection, cleaning, and validation. The eCRFs will include programmable edits to obtain immediate feedback if data are missing, out of range, illogical, or potentially erroneous. Concurrent manual data review will be performed based on parameters dictated by the plan. Ad hoc queries will be generated within the electronic data capture (EDC) system and followed up until resolution.

High data quality standards will be maintained, and processes and procedures will be utilized to repeatedly ensure that the data are as clean and accurate as possible when presented analysis.

Data quality will be enhanced through a series of programmed data quality checks that automatically detect out-of-range or anomalous data.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years of age at the time of signing the informed consent form.
2. Subject has biopsy-proven malignancy and is starting myelosuppressive chemotherapy in the neoadjuvant/adjuvant or first line advanced/metastatic setting with at least 4 anticipated chemotherapy cycles.
3. Subject's life expectancy > 6 months.
4. Subject is in a high-risk category for FN: 1) the subject is starting or has, within the past 7 days, started a myelosuppressive chemotherapy regimen with a high (> 20%) FN risk 2) patient is on a chemotherapy regimen with an intermediate (10-20%) FN risk but is determined by his or her treating physician to be at a high-risk (therefore requiring primary prophylaxis with myeloid growth factor), or 3) patient is on secondary prophylaxis for FN (per NCCN guidelines).
5. Subject is starting adjuvant chemotherapy, neoadjuvant chemotherapy, or first line chemotherapy in the metastatic setting and will be receiving at least 4 cycles of planned chemotherapy.
6. Subjects already receiving any other Pegfilgrastim (switching) as a FN prophylaxis will be allowed to enroll so long as they have at least two cycles left in their planned treatment.

Exclusion Criteria:

1. Subject initiating chemotherapy regiment wtih <14 days between cytotoxic and G-CSF drug dosing.
2. Planned chemotherapy dose reduction for cycle 1.
3. Known history of serious allergic reactions to Pegfilgrastim or Filgrastim.
4. Contraindication to short acting G-CSFs, Pegfilgrastim biosimilar PFS
5. Currently receiving treatment in another investigational device or drug study, or

   ≤ 28 days before screening/enrollment since ending treatment on another investigational device or drug study.
6. Subject who has received radiation < 2 weeks prior to study enrollment.
7. Any co-morbidity in the opinion of the investigator that will prevent the subject from receiving chemotherapy.
8. Subject has significant abnormalities on the most recent laboratory test prior to Screening/Enrollment per the Investigator including but not limited to the following:

   white blood cell (WBC) < 4, ANC < lower limit of normal (LLN), hemoglobin < 10 g/dL, hematocrit < 30%, platelet count < 100,000, creatinine ≥ 1.5 or glomerular filtration rate < 30 (as calculated by Cockcroft-Gault Equation), total bilirubin ≥ 2.0, aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≥ 3 x upper limit of normal (ULN), subject without liver metastasis or AST/ALT ≥ 5 ULN in a subject with liver metastasis
9. Known human immunodeficiency virus (HIV) infection by history.
10. History of solid organ or stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will comprise of individuals with biopsy-verified cancer who are receiving myelosuppressive chemotherapies and who have been prescribed Udenyca due to their high risk of febrile neutropenia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of FN in real-world outcome setting | 24 months
  Calculation of the incidence of FN (as defined by NCCN) among subjects in a real-world outcome setting who are 1) being treated with myelosuppressive chemotherapy for the treatment of non- myeloid malignancies and 2) receiving Udenyca with every administered chemotherapy cycle for FN prophylaxis.

SECONDARY OUTCOMES:
The incidence of FN in a curative setting | 24 months
  Calculation of the incidence of FN (as defined by NCCN) among subjects in a curative setting who are 1) being treated with myelosuppressive chemotherapy for the treatment of non-myeloid malignancies and 2) receiving Udenyca with every administered chemotherapy cycle for FN prophylaxis
The incidence in FN in a palliative setting | 24 months
  Calculation of the incidence of FN (as defined by NCCN) among subjects in a palliative setting who are 1) being treated with myelosuppressive chemotherapy for the treatment of non-myeloid malignancies and 2) receiving Udenyca with every administered chemotherapy cycle for FN prophylaxis.
Measure quality of life in subjects receiving Udenyca for FN prophylaxis | 24 months
  Measurement of HRQoL in subjects who received Udenyca with FN prophylaxis
To compare the incidence of FN in subjects who switched to Udenyca | 24 months
  To compare the incidence of FN in subject who switched to Udenyca with the estimated incidence of FN in subjects who received other Pegfilgrastims for FN prophylaxis (overall) in curative and palliative settings.

CONTACTS AND LOCATIONS:
Overall Officials: Sashi Naidu, MD, Principal Investigator — Carolina Blood and Cancer Care
Locations (3):
- United States (3):
  - Southern Oncology Specialists, Charlotte, North Carolina
  - Coastal Cancer Center, Myrtle Beach, South Carolina
  - Carolina Blood and Cancer Care, PA, Rock Hill, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided